CLINICAL TRIAL: NCT00345787
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Determine the Efficacy and Safety of BTDS Compared to Placebo in Subjects With Moderate to Severe Osteoarthritic Pain of the Hip or Knee
Brief Title: Comparison of BTDS (Buprenorphine Transdermal System) and Placebo in Osteoarthritic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma K.K. (Industry)
Responsible Party: Mutsukuni Kataoka, Mundipharma K.K.
Organization: Mundipharma Pte Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUP3801
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Pain; Osteoarthritis
Keywords: Osteoarthritic Pain
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 0 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental)
  Interventions: Drug: Buprenorphine Transdermal System

INTERVENTIONS:
Drug: Placebo — Corresponding placebo is applied for 12weeks
  Arms: 0
Drug: Buprenorphine Transdermal System — Buprenorphine Transdermal System 5, 10 or 20mg/patch is applied for 12weeks
  Arms: 1

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of BTDS compared to placebo in subjects with moderate to severe osteoarthritic pain of the hip or knee.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy and safety of buprenorphine transdermal system (BTDS) compared to placebo in subjects with moderate to severe osteoarthritic pain of the hip or knee who have a sub-optimal response to their non-opioid analgesic treatment and require opioid analgesics for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ages 40 years or older.
* Clinical diagnosis of osteoarthritis (OA) of the hip or knee.

Exclusion Criteria:

* Subjects who have a current or past history of chronic disease(s), in addition to OA, requiring frequent analgesic therapy (e.g. headache, fibromyalgia, gout, rheumatoid arthritis, low back pain, and diabetic neuropathy).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2006-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The time to the development of inadequate analgesia | Up to 12weeks

SECONDARY OUTCOMES:
Percentage of subjects who developed inadequate analgesia, 'Average pain over the last 24 hours' scores | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mutsukuni Kataoka, Study Chair — Department Head, Clinical Trial Operations, Clinical Development, Mundipharma K.K.
Locations (28):
- Japan (28):
  - Investigational Site, Nagoya, Aichi-ken
  - Investigational Site, Okazaki, Aichi-ken
  - Investigational Site, Ichikawa, Chiba
  - Investigational Site, Matsudo, Chiba
  - Investigational Site, Nagareyama, Chiba
  - Investigational Site, Fukui-shi, Fukui
  - Investigational Site, Annaka, Gunma
  - Investigational Site, Takasaki, Gunma
  - Investigational Site, Chitose, Hokkaido
  - Investigational Site, Sapporo, Hokkaido
  - Investigational Site, Kako, Hyōgo
  - Investigational Site, Kobe, Hyōgo
  - Investigational Site, Yokohama, Kanagawa
  - Investigational Site, Jōyō, Kyoto
  - Investigational Site, Sendai, Miyagi
  - Investigational Site, Isahaya, Nagasaki
  - Investigational Site, Osaka, Osaka
  - Investigational Site, Kasukabe, Saitama
  - Investigational Site, Koshigaya, Saitama
  - Investigational Site, Hikone, Shiga
  - Investigational Site, Adachi City, Tokyo
  - Investigational Site, Arakawa City, Tokyo
  - Investigational Site, Edogawa City, Tokyo
  - Investigational Site, Koto, Tokyo
  - Investigational Site, Setagaya City, Tokyo
  - Investigational Site, Suginami, Tokyo
  - Investigational Site, Himi, Toyama
  - Investigational Site, Kurobe-shi, Toyama